CLINICAL TRIAL: NCT04591535
Title: An Open Label, Balanced, Randomised, Four-treatment, Four-period, Four-sequence, Single Oral Dose, Crossover PK Study of WD-1603 in Normal, Healthy, Adult Human Subjects Under Fed Conditions
Brief Title: PK Study of WD-1603 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong WD Pharmaceutical Co., Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WD-1603-1003
Record Dates: First submitted 2020-09-11; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- WD-1603 (tablet strength 1) single dose (Experimental): A single oral dose of carbidopa/levodopa extended release tablets (WD-1603 tablet strength 1) will be administered to each subject within 5 minutes at 30 minutes after serving standardized vegetarian breakfast under fed condition in each period as per randomization schedule.
  Interventions: Drug: WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS
- WD-1603 (tablet strength 2) single dose (Experimental): A single oral dose of carbidopa/levodopa extended release tablets (WD-1603 tablet strength 2) will be administered to each subject within 5 minutes at 30 minutes after serving standardized vegetarian breakfast under fed condition in each period as per randomization schedule.
  Interventions: Drug: WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS
- WD-1603 (tablet strength 3) single dose (Experimental): A single oral dose of carbidopa/levodopa extended release tablets (WD-1603 tablet strength 3) will be administered to each subject within 5 minutes at 30 minutes after serving standardized vegetarian breakfast under fed condition in each period as per randomization schedule.
  Interventions: Drug: WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS
- WD-1603 (tablet strength 4) single dose (Experimental): A single oral dose of carbidopa/levodopa extended release tablets (WD-1603 tablet strength 4) will be administered to each subject within 5 minutes at 30 minutes after serving standardized vegetarian breakfast under fed condition in each period as per randomization schedule.
  Interventions: Drug: WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS

INTERVENTIONS:
Drug: WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS — WD-1603 CARBIDOPA/LEVODOPA EXTENDED-RELEASE TABLETS
  Other Names: WD-1603

SUMMARY:
An open label, balanced, randomised, four-treatment, four-period, four-sequence, single oral dose, crossover Pharmacokinetics study of WD-1603 carbidopa/levodopa extended-release tablets in normal, healthy, adult human subjects under fed conditions. A single oral dose of (either Treatment A or B or C or D) carbidopa/levodopa extended release tablets will be administered to each subject within 5 minutes after completion of standardized vegetarian breakfast under fed condition in each period as per randomization schedule.

DETAILED DESCRIPTION:
This is an open label, balanced, randomised, four-treatment, four-period, four-sequence, single oral dose, crossover Pharmacokinetics study of WD-1603 carbidopa/levodopa extended-release tablets in normal, healthy, adult human subjects under fed conditions. A single oral dose of (either Treatment A or B or C or D) carbidopa/levodopa extended release tablets will be administered to each subject within 5 minutes after completion of standardized vegetarian breakfast under fed condition in each period as per randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy adult human volunteers between 18 to 45 years of age (both inclusive).
2. Having a Body Mass Index (BMI) between 18.5 to 29.9 (both inclusive), calculated as weight in kg / height in m2, a minimum body weight of 50.0 kg.
3. Not having any significant disease or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12- lead ECG and X-ray chest (P/A view) recordings.
4. Able to understand and comply with the study procedures, in the opinion of the principal investigator.
5. Able to give voluntary written informed consent for participation in the trial.
6. In case of female subjects:

a. Surgically sterilized at least 6 months prior to study participation or If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And b. Serum Pregnancy test must be negative.

g.Female must also be willing to abstain from ovum donation from Screening and for at least 28 days after the last study drug administration.

h.Female subjects of non-childbearing potential must be either post-menopausal (post-menopausal is defined as being amenorrheic for at least 1 year without another cause and a follicle-stimulating hormone [FSH] level ≥26 IU/L) or surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).

i.Male subjects with female sexual partners of childbearing potential must be willing to use and willing to continue using medically acceptable contraception (true abstinence, vasectomy, or male condom for subjects plus an additional method of contraception for their female partners) from dosing until 28 days following the last administration of study drug.

j.Men must also be willing to abstain from sperm donation from Screening and for at least 28 days after the last study drug administration.

k.Subjects should be literate.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to Carbidopa or Levodopa or any of the excipients or any related drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, cardiovascular, immunological, dermatological, gastrointestinal system, and central nervous system with dyskinesia, depression, suicidal thought, or any other body system.
3. History or presence of ophthalmic diseases such as wide angle glaucoma and ocular hypertension.
4. Ingestion of a medicine (prescribed & over the counter (OTC) medication including herbal remedies and MAO inhibitors) at any time within 30 days before dosing in Period I. In any such case subject selection will be at the discretion of the Principal Investigator.
5. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
6. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.

g.A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to dosing in Period I.

h.Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study.

i.The presence of clinically significant abnormal laboratory values during screening.

j.History or presence of psychiatric disorders. k.A history of difficulty in donating blood. l.Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.

m.Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.

* If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.

  n.A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.

  o.A positive test result for HIV (1 &/or 2) antibody. p.An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine in period I. In any such case subject selection will be at the discretion of the Principal Investigator.

  q.Consumption of grapefruit or grapefruit products within 72 hours prior to dosing in period-I.

  r.Difficulty in swallowing oral solid dosage form like tablets or capsules. s.Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 2
  the maximum plasma concentrations
AUC | Day 1 and Day 2
  areas under the plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Shrikrishna Kolte, Doctor, Principal Investigator — Lambda Therapeutic Research Limited, Ahmedabad,India
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, India